CLINICAL TRIAL: NCT01262092
Title: Effects of Gabapentin Versus Placebo on Buprenorphine Detoxification of Opioid-dependent Individuals
Acronym: Detox
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01-DA010017-pilot; 112714 (Other: UAMS IRB); R01DA010017 (NIH)
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Results first posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Opioid Dependence; Opioid Withdrawal; Opioid Detoxification
Keywords: opioid dependent; detoxification; buprenorphine; suboxone; opiate
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Gabapentin; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Active Comparator): Buprenorphine will be given along with 2 capsules of gabapentin in the morning and 2 take-home capsules of gabapentin for night.
  Interventions: Drug: Buprenorphine
- Placebo (Placebo Comparator): Buprenorphine will be given, with 2 capsules of placebo in the morning and 2 take-home capsules of placebo in the evening
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Induction onto buprenorphine to a stable dose of 12mg/day. Then induction onto either 0 or 1600mg of gabapentin. Once the maintenance dose of gabapentin is reached a 10-day buprenorphine detoxification will begin.
  Other Names: Neurontin, Suboxone,

SUMMARY:
This study involves inducting treatment seeking opioid dependent participants onto buprenorphine. Once the participant reaches a stable dose they will receive either placebo or gabapentin to determine if gabapentin helps ease withdrawal symptoms while the participant undergoes a 10-day buprenorphine detoxification.

ELIGIBILITY:
Inclusion Criteria:

* Availability to attend clinic 6 days a week for approximately 30-60 minutes.
* Participants must fulfill DSM-IV criteria for opioid dependence. These criteria will be ascertained in the following manner: the physician will determine whether the individual is appropriate based on several clinical assessments that are routinely employed by methadone program physicians, including history and severity of opioid use, presence of track marks, prior treatment history, self-reported and/or observed signs and symptoms of opioid withdrawal. If any individual's degree of opioid dependence is questionable, that person will be excluded from further consideration as a participant.
* Participants must submit a urine negative for drugs of abuse other than opioids prior to starting the study.

Exclusion Criteria:

* Unstable medical condition or stable medical condition that would interact with study medications or participation.
* History of major psychiatric disorder (psychosis, schizophrenia, bipolar, depression)
* Pregnancy or plans to become pregnant or inadequate birth control (adequate birth control includes abstinence, condoms, birth control pills, etc).
* Present or recent use of over-the-counter psychoactive drug, prescription psychoactive drug or drug (including Maalox) that would have major interaction with drugs to be tested.
* Liver function tests greater than 3 times normal, BUN and Creatinine outside normal range, or thyroid function tests outside normal range.
* EKG abnormalities including but not limited to: bradycardia (<60 bpm); prolonged QTc interval (>450 msec); Wolff-Parkinson White syndrome; wide complex tachycardia; 2nd degree, Mobitz type II heart block; 3rd degree heart block; left or right bundle branch block.
* Physical dependence on alcohol or drugs other than opioids or tobacco (as determined by physician assessment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, Ph.D., Principal Investigator — UAMS Center for Addiction Research
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty treatment-seeking opioid-dependent individuals were recruited from Central Arkansas by ads, word-of-mouth and referrals in October 2010 and January 2011-December of 2011. An experienced research staff member obtained informed consent interviewed subjects in a private office on the 4th floor of the Psychiatric Research Institute.
Pre-assignment Details: On Tuesday of Week 1, participants were randomized into treatment groups based on withdrawal symptoms score, sex and primary opioid of abuse using an urn randomization procedure. This was done to ensure that groups are balanced with respect to potential prognostic factors.
Period: Buprenorphine+Gabapentin/Plac Induction
Arm/Group | Gabapentin | Placebo
Started | 16 | 14
Completed | 13 | 13
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 1 | 0
Period: Buprenorphine Taper
Arm/Group | Gabapentin | Placebo
Started | 12 (One left the study prior to starting the taper due to pharmacy error (started taper in wk 2)) | 13
Completed | 11 | 12
Not Completed | 1 | 1
Not completed — noncompliance - missed medication | 1 | 1
Period: Gabapentin Taper
Arm/Group | Gabapentin | Placebo
Started | 10 (One participant dropped out after the buprenorphine taper but prior to the gabapentin taper) | 11 (One participant dropped out after the buprenorphine taper but prior to the gabapentin taper)
Completed | 9 | 11
Not Completed | 1 | 0
Not completed — noncompliance - missed medications | 1 | 0

BASELINE CHARACTERISTICS:
Population: analysis was based on those starting the buprenorphine detox except for one subject in the gabapentin arm (evidence of noncompliance with medication procedures and diversion)
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.00 (11.05) | 30.31 (10.62) | 29.71 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Illicit Opioid Use as Determine by Urine Dipsticks
Description: urine data are from those obtained during the buprenorphine taper
Time Frame: 3x weekly during wks 3 and 4
Population: Those who started the bup detox (N=24) excluding 1 subjects' data in the gabapentin group due to evidence of noncompliance with medication procedures and diversion (N=1).
Measure: Mean (Standard Error); unit: % of urines positive for opioids
Units Other Than Participants: urine samples
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 11 | 13
Number analyzed (urine samples) | 65 | 75
% of urines positive for opioids | 13.64 (5.69) | 32.56 (9.93)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; test null hypothesis that gbp and pla did not differ in terms of opioid-positive urines during the buprenorphine detox. For the analysis, data from 2 participants in the GBP groups were excluded due to evidence of medication diversion (N=1) and not being maintained on the 1600 mg/day dose of GBP (N=1); Test type: Superiority or Other; p = 0.035, Mixed Models Analysis — p values <0.05 considered statistically significant; Used proc GLIMMIX to model group by time (6 study visits); Mean Difference (Final Values) = -8.2887

ADVERSE EVENTS:
Arm/Group | Gabapentin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 10/16 | 4/14
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=16) | Placebo (N=14)
Dizziness/Lightheadedness (Nervous system disorders) | 1 (1) | 2 (2)
nausea/vomiting (Gastrointestinal disorders) | 4 (4) | 2 (3)
Sleepiness/Fatigue/Somnulence (Psychiatric disorders) | 3 (3) | 1 (1)
Vivid, disturbing dreams, nightmares (Psychiatric disorders) | 4 (4) | 0 (0)
muscle twitches/cramps (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes